CLINICAL TRIAL: NCT05600569
Title: Registry of the Spanish Society of Thoracic Surgery (ReSECT)
Brief Title: Registry of the Spanish Society of Thoracic Surgery
Acronym: ReSECT
Status: Recruiting | Type: Observational
Sponsor: Sociedad Española de Cirugía Torácica (Other)
Responsible Party: Sponsor
Other Study IDs: sect/resect/01
Record Dates: First submitted 2022-10-19; First posted 2022-10-31 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Surgical Procedures; Thoracic Surgery, Video-assisted; Robotic Surgical Procedures; Thoracotomy; Lung Neoplasm
Keywords: Pneumonectomy; Lobectomy; Segmentectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All the target population: Patients who will undergo any surgical procedure in a Spanish Thoracic Surgery Department

SUMMARY:
ReSECT is a project promoted by the Spanish Society of Thoracic Surgery with the aim not only to become an indefinite, dynamic and inclusive registry, but also to establish a common structural framework for the development of future multicentre projects in the field of thoracic surgery in Spain.

The goal of this nationwide prospective observational registry is:

* To develop and validate forecasting tools based on powerful computational methods with the goal of assisting in decision-making and improving quality of care.
* To evaluate the progressive implementation of certain surgical techniques that are on the rise, new technologies and future health programs.
* To be aware of our results as specialty and professionals and to serve as a permanent benchmarking instrument in thoracic surgery.

The first part of ReSECT, based on a personal registry design, will contemplate any thoracic surgical procedure performed by thoracic surgeons and residents in thoracic surgery in our country. Additionally, the Spanish thoracic surgery departments that voluntarily accept to collectively participate will contribute to specific surgical processes focused on certain procedures with specific objectives to be progressively implemented.

The first and only surgical process implemented since the start of the ReSECT project will focus on patients to undergo anatomical lung resection with special interest in those cases whose reason for intervention was lung cancer.

The main questions to answer in case of that first surgical process include:

* What is the performance of current predictive models for perioperative and oncological outcomes in our country?
* How could we modify previous predictive models to improve their performance?
* What is the implementation of current guideline recommendations in our country and across institutions?
* What is the potential impact of deviations from current recommendations?
* What is my performance compared to the rest of the thoracic surgical departments in my country in terms of perioperative and oncological outcomes?

ReSECT does not consider prespecified comparison groups of patients.

DETAILED DESCRIPTION:
ReSECT is intended for SECT members including thoracic surgery specialists and residents with professional practice in Spain, as well as thoracic surgery departments in our country.

Participation in ReSECT may be at the individual level (personal surgical registry) or by department (ReSECT surgical processes). Those thoracic surgery departments interested in participating in a surgical process implemented in ReSECT must be represented by a single responsible hospital user.

ReSECT will be a clinical registry based on surgical procedures. The retrospective and prospective nature of the personal surgical record will be determined by the user's ability to include records of patients who underwent surgery prior to the approval of the current project. However, the "retrospective patients" to be included must belong to the centre associated with each user at the time of registering on the platform. In other words, it will not be feasible to include patients operated on in other institutions where the professional had previously worked.

The first ReSECT surgical process about anatomical lung resections and the successive processes that are to be created in the future, will only contemplate patients operated on prospectively with respect to the date of approval of each surgical process.

ELIGIBILITY:
The inclusion criteria will depend on the section of the registry to be considered.

* Personal registry: patients undergoing any type of surgical intervention.
* Registry of surgical processes by departments: patients undergoing an anatomical pulmonary resection as the first process to be implemented at the time ReSECT is to be established.

Exclusion Criteria:

* Patients who could reject to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients that could requiere an intervention in the Spanish Thoracic Surgery Departments
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of perioperative mortality | From surgery date to hospital discharge day or within ninety days.
  Mortality during hospitalization or that occurred within thirty and ninety days after surgery.
Rate and severity of perioperative morbidity | From surgery date to hospital discharge day or within thirty days.
  Complications occurred during hospitalization will be classified into 3 groups: cardiovascular, respiratory and other type of complications. Each of these groups of complications will be classified based on the most severe specific complication according to the Clavien-Dindo classification (grade I, II, IIIa, IIIb, IVa, IVb, V).
  Specific respiratory complications: initial ventilator support > 48h, re-intubation, ARDS, pneumonia, atelectasis, air leak > 5 days, pulmonary embolism, acute respiratory failure, phrenic palsy, pulmonary infarction, pneumothorax, pleural effusion, subcutaneous emphysema, chylothorax, bronchopleural fistula, others.
  Specific cardiovascular complications: blood transfusion, arrhythmia, myocardial infarction, heart failure, cerebrovascular accident, deep vein thrombosis, others.
  Other type of complications: no-respiratory sepsis, wound infection, renal failure, delirium, others.
Overall survival | Five-year follow-up after surgery
  Overall survival after anatomical resection for lung cancer. The outcome will include exitus for any reason.
Disease specific survival | Five-year follow-up after surgery
  Disease free survival after anatomical resection for lung cancer. The outcome will include exitus for lung cancer progesssion.
Recurrence free survival | Five-year follow-up after surgery.
  Recurrence free survival after anatomical resection for lung cancer. The outcome will include recurrence of lung cancer.

SECONDARY OUTCOMES:
Rate of hospital readmission | From hospital discharge day to thirty days afterwards.
  Readmissions within thirty days of discharge from hospital for reasons related to the surgical procedure.
Diagnosis and severity of complications during hospital readmission. | From hospital readmission date to hospital discharge day or within 30 days
  Primary reason for readmission and severity of complications from readmission date to hospital discharge day
Unplanned Intensive Care | From day of surgery to day of hospital discharge or within 30 days
  Rate of patients who required unplanned intensive care unit admission
Rate of patients that required surgical reintervention | From surgery date to hospital discharge day and from hospital readmission date to hospital discharge day or within 30 days
  Surgical reinterventions will be considered when related to complications secondary to the main surgical procedure.
  This rate will be calculated: number of patients that required reintervention during main hospitalization of after readmission / total number of patients.
Rate of patients with functional status classified as independent, partially independent of totally dependent | The day of hospital discharge or within 30 days after surgery.
  Functional status will be referred to patient ability to perform basic and instrumental activities of daily living.
  Patients will be classified into:
  1. Independent: autonomous patient to carry out most of the instrumental activities of daily living (pet care, raising kids, use of communication systems, mobility in the community, management of financial issues, health care and support, maintain a home, food preparation and cleaning, security procedures and emergency responses, go shopping).
  2. Partially dependent: autonomous patient for most of the basic activities of daily living (bath / shower, locker room, feeding, sphincters control, functional mobility, care of personal technical aids, personal hygiene and grooming, sexual activity, go sleeping, toilet hygiene), but unable to perform most instrumental activities of daily living.
  3. Totally dependent: patient who requires help to carry out most of the basic activities of daily living.
Rate of patients with invasive mediastinal staging | From three months before surgery to surgical intervention date
  Number of patients with diagnosis of lung cancer who underwent invasive staging of the mediastinum / number of patients with lung cancer who meet criteria for invasive staging of the mediastinum according to current guidelines.
Rate of complete resection for lung cancer | During the surgery
  Number of patients with lung cancer who underwent complete resection / number of patients with lung cancer who underwent surgical resection.
Distribution of patients according to type of lymphadenectomy | During the surgery
  Patients operated on for lung cancer will be classified according to type of lymphadenectomy performed into:
  1. Minor Lymphadenectomy.
  2. Lobe-specific systematic lymph node dissection: exeresis of the mediastinal tissue that contains the lymph nodes of certain lymph node stations is performed, depending on the location of the tumor.
     * Tumor in the right upper lobe or middle lobe: 2R, 4R and 7.
     * Tumor in the lower right lobe: 4R, 7, 8 and 9.
     * Tumor in the upper left lobe: 5, 6 and 7.
     * Tumor in the lower left lobe: 7, 8 and 9.
  3. Systematic lymph node dissection: dissection and exeresis of the mediastinal tissue that contains the lymph nodes following the anatomical limits. It is recommended that at least 3 mediastinal lymph node stations be excised, always including the subcarinal, in addition to the hilar and intrapulmonary stations.
Rate of occult pN2 disease | During the surgery
  Number of patients operated on for lung cancer with pathological N2 disease and clinical N0-N1 disease / Number of patients operated on for lung cancer with clinical N0-N1 disease.
Mean postoperative stay | From day of surgery to day of hospital discharge or within 3 months.
  Number of days of hospitalization after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raúl Embún, PhD, Study Director — Hospital Universitario Miguel Servet / raulembun@gmail.com / Phone: +34 635 492179
Locations (1):
- Hospital Universitario Miguel Servet. Hospital Clínico Universitario Lozano Blesa. IIS Aragón. Universidad Zaragoza., Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Embun R, Royo-Crespo I, Recuero Diaz JL, Bolufer S, Call S, Congregado M, Gomez-de Antonio D, Jimenez MF, Moreno-Mata N, Aguinagalde B, Amor-Alonso S, Arraras MJ, Blanco Orozco AI, Boada M, Cabanero Sanchez A, Cal Vazquez I, Cilleruelo Ramos A, Crowley Carrasco S, Fernandez-Martin E, Garcia-Barajas S, Garcia-Jimenez MD, Garcia-Prim JM, Garcia-Salcedo JA, Gelbenzu-Zazpe JJ, Giraldo-Ospina CF, Gomez Hernandez MT, Hernandez J, Wolf JDI, Jauregui Abularach A, Jimenez U, Lopez Sanz I, Martinez-Hernandez NJ, Martinez-Tellez E, Milla Collado L, Mongil Poce R, Moradiellos-Diez FJ, Moreno-Balsalobre R, Moreno Merino SB, Obiols C, Quero-Valenzuela F, Ramirez-Gil ME, Ramos-Izquierdo R, Rivo E, Rodriguez-Fuster A, Rojo-Marcos R, Sanchez-Lorente D, Sanchez Moreno L, Simon C, Trujillo-Reyes JC, Hernando Trancho F. Spanish Video-Assisted Thoracic Surgery Group: Method, Auditing, and Initial Results From a National Prospective Cohort of Patients Receiving Anatomical Lung Resections. Arch Bronconeumol. 2020 Nov;56(11):718-724. doi: 10.1016/j.arbr.2020.01.009. PMID 35579917
- [Background] Gomez de Antonio D, Crowley Carrasco S, Romero Roman A, Royuela A, Sanchez Calle A, Obiols Fornell C, Call S, Embun R, Royo I, Recuero JL, Cabanero A, Moreno N, Bolufer S, Congregado M, Jimenez MF, Aguinagalde B, Amor-Alonso S, Arraras MJ, Blanco Orozco AI, Boada M, Cal I, Cilleruelo Ramos A, Fernandez-Martin E, Garcia-Barajas S, Garcia-Jimenez MD, Garcia-Prim JM, Garcia-Salcedo JA, Gelbenzu-Zazpe JJ, Giraldo-Ospina CF, Gomez Hernandez MT, Hernandez J, Illana Wolf JD, Jauregui Abularach A, Jimenez U, Lopez Sanz I, Martinez-Hernandez NJ, Martinez-Tellez E, Milla Collado L, Mongil Poce R, Moradiellos-Diez FJ, Moreno-Basalobre R, Moreno Merino SB, Quero-Valenzuela F, Ramirez-Gil ME, Ramos-Izquierdo R, Rivo E, Rodriguez-Fuster A, Rojo-Marcos R, Sanchez-Lorente D, Moreno LS, Simon C, Trujillo-Reyes JC, Lopez Garcia C, Fibla Alfara JJ, Sesma Romero J, Hernando Trancho F. Surgical Risk Following Anatomic Lung Resection in Thoracic Surgery: A Prediction Model Derived from a Spanish Multicenter Database. Arch Bronconeumol. 2022 May;58(5):398-405. doi: 10.1016/j.arbres.2021.01.037. Epub 2021 Feb 24. English, Spanish. PMID 33752924
- [Background] Aguinagalde B, Insausti A, Lopez I, Sanchez L, Bolufer S, Embun R; en representacion del Grupo Espanol de Cirugia Toracica Video-asistida. VATS lobectomy morbidity and mortality is lower in patients with the same ppoDLCO: Analysis of the database of the Spanish Video-Assisted Thoracic Surgery Group. Arch Bronconeumol. 2021 Dec;57(12):750-756. doi: 10.1016/j.arbr.2021.10.005. Epub 2021 Oct 30. PMID 35698981
- [Background] Gomez Hernandez MT, Novoa Valentin NM, Fuentes Gago MG, Embun Flor R, Gomez de Antonio D, Jimenez Lopez MF; Spanish Group of Video-assisted Thoracic Surgery. Predictive factors of pathological complete response after induction (ypT0N0M0) in non-small cell lung cancer and short-term outcomes: Results of the Spanish Group of Video-assisted Thoracic Surgery (GE-VATS). Cir Esp (Engl Ed). 2022 Jun;100(6):345-351. doi: 10.1016/j.cireng.2022.05.025. Epub 2022 May 25. PMID 35643356
- [Background] Gomez Hernandez MT, Novoa Valentin NM, Embun Flor R, Varela Simo G, Jimenez Lopez MF; Grupo Espanol de Cirugia Toracica Videoasistida (GEVATS). Predictive factors of prolonged postoperative length of stay after anatomic pulmonary resection. Cir Esp (Engl Ed). 2023 Jan;101(1):43-50. doi: 10.1016/j.cireng.2022.06.048. Epub 2022 Jul 3. PMID 35787477
- [Background] Obiols C, Call S, Rami-Porta R, Jaen A, Gomez de Antonio D, Crowley Carrasco S, Royo-Crespo I, Embun R. Radicality of lymphadenectomy in lung cancer resections by thoracotomy and video-assisted thoracoscopic approach: A prospective, multicentre and propensity-score adjusted study. Lung Cancer. 2022 Mar;165:63-70. doi: 10.1016/j.lungcan.2022.01.004. Epub 2022 Jan 7. PMID 35091211
- [Background] Sesma J, Bolufer S, Garcia-Valentin A, Embun R, Lopez IJ, Moreno-Mata N, Jimenez U, Trancho FH, Martin-Ucar AE, Gallar J; Spanish Video-Assisted Thoracic Surgery Group. Thoracoscopic segmentectomy versus lobectomy: A propensity score-matched analysis. JTCVS Open. 2022 Jan 22;9:268-278. doi: 10.1016/j.xjon.2022.01.009. eCollection 2022 Mar. PMID 36003470
- [Background] Lopez I, Aguinagalde B, Urreta I, Royo I, Bolufer S, Sanchez L, Zabaleta J, Fernandez-Monge A, Recuero-Diaz JL, Sesma J, Amor S, Moradiellos FJ, Arraras MJ, Blanco AI, Boada M, Sanchez D, Cabanero A, Moreno N, Cal I, Moreno R, Cilleruelo A, Crowley S, Gomez D, Fernandez E, Hernando F, Garcia S, Lopez C, Garcia MD, Garcia JM, Rivo JE, Garcia JA, Gelbenzu JJ, Ramirez ME, Giraldo CF, Mongil R, Gomez MT, Jimenez M, Henandez J, Fibla JJ, Illana JD, Jauregui A, Jimenez U, Rojo R, Martinez NJ, Martinez E, Trujillo JC, Milla L, Moreno SB, Congregado M, Obiols C, Call S, Quero F, Ramos R, Rodriguez A, Simon CM, Embun R. Results in mediastinal lymph node staging of surgical lung cancer: Data from the prospective cohort of the Spanish Video-Assisted Thoracic Surgery Group. Cir Esp (Engl Ed). 2023 Jun;101(6):408-416. doi: 10.1016/j.cireng.2022.06.006. Epub 2022 Jun 6. PMID 35671974
- [Background] Gomez de Antonio D, Crowley Carrasco S, Romero Roman A, Royuela A, Gil Barturen M, Obiols C, Call S, Royo I, Recuero JL, Cabanero A, Moreno N, Embun R; Spanish Group of Video Assisted Thoracic Surgery (GEVATS). External validation of the European Society of Thoracic Surgeons morbidity and mortality risk models. Eur J Cardiothorac Surg. 2022 Aug 3;62(3):ezac170. doi: 10.1093/ejcts/ezac170. PMID 35301527
- [Background] Pons A, Guirao A, Fibla JJ, Carvajal C, Embun R, Sanchez D, Gevats, Hernandez J. National evaluation of risk factors for unplanned readmission after lung resection. Eur J Cardiothorac Surg. 2022 May 27;61(6):1251-1257. doi: 10.1093/ejcts/ezac081. PMID 35218337
- [Background] Recuero-Diaz JL, Royo-Crespo I, Gomez de-Antonio D, Call S, Aguinagalde B, Gomez-Hernandez MT, Hernandez-Ferrandez J, Sanchez-Lorente D, Sesma-Romero J, Rivo E, Moreno-Mata N, Embun R. Treatment and intention-to-treat propensity score analysis to evaluate the impact of video-assisted thoracic surgery on 90-day mortality after anatomical resection for lung cancer. Eur J Cardiothorac Surg. 2022 Aug 3;62(3):ezac122. doi: 10.1093/ejcts/ezac122. PMID 35213711
- [Background] Cabanero Sanchez A, Munoz Molina GM, Fra Fernandez S, Muriel Garcia A, Cilleruelo Ramos A, Martinez Hernandez N, Hernando Trancho F, Moreno Mata N; GE-VATS. Impact of neoadjuvant therapy on postoperative complications in non-small-cell lung cancer patients subjected to anatomic lung resection. Eur J Surg Oncol. 2022 Sep;48(9):1947-1953. doi: 10.1016/j.ejso.2022.03.008. Epub 2022 Mar 29. PMID 35379545
- See also: Spanish Society of Thoracic Surgery — https://www.sect.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT05600569/Prot_SAP_ICF_000.pdf